CLINICAL TRIAL: NCT03720704
Title: Post-Market Registry of the GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis Implanted in Peripheral Vessels
Acronym: EXPAND
Status: Active, not recruiting | Type: Observational
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Other Study IDs: VBX 17-04
Record Dates: First submitted 2018-09-14; First posted 2018-10-25 (Actual); Results first posted 2024-02-16 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Peripheral Vascular Diseases
Keywords: Lesion-exclusion; Visceral Perfusion; Luminal Reconstruction; Occlusive Disease
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- GORE VIABAHN VBX Balloon Expandable Endoprosthesis: The GORE VIABAHN VBX Balloon Expandable Endoprosthesis will be implanted according to the institution standard of practice in patients needing preservation of peripheral vessels due to multiple pathologies and conditions.
  Interventions: Device: GORE VIABAHN VBX Balloon Expandable Endoprosthesis

INTERVENTIONS:
Device: GORE VIABAHN VBX Balloon Expandable Endoprosthesis — GORE VIABAHN VBX Balloon Expandable Endoprosthesis will be implanted in peripheral vessels in patients who require interventional treatment.

SUMMARY:
The primary objective of the VBX 17-04 registry is to collect post-market safety and performance data of the GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis (VBX Stent Graft) in peripheral vessels in patients who require interventional treatment

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Signed informed consent form
* Endovascular indication for treatment based on treating physician's best medical judgment.
* Intend for no other stents to be placed in the same peripheral vessel(s) targeted for VBX Stent Graft placement.
* Willingness of the patient to adhere to standard of care follow-up requirements.

Exclusion Criteria:

* Known hypersensitivity to heparin or a previous incident of Heparin-Induced Thrombocytopenia (HIT) type II.
* Participation in concurrent research study or registry which may confound registry results, unless approved by Gore.
* Pregnant or breast-feeding female at time of informed consent signature.
* Life expectancy < 12 months due to comorbidities.
* Use of the VBX Stent Graft is for the treatment of de novo iliac occlusive disease.
* Use of the VBX Stent Graft is for the treatment of aortic coarctations.
* Use of the VBX Stent Graft in the coronary, pulmonary, carotid, vertebral, isolated infrarenal aortic, or vena cava vessels.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry has been designed with broad eligibility criteria to capture real-world VBX Stent Graft use, in multiple pathologies and in conditions needing preservation of peripheral vessels.
Sampling Method: Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2027-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Gargiulo, MD, Principal Investigator — Azienda Ospedaliera Policlinico Sant'Orsola Malpighi
Locations (11):
- Hôpital Marie Lannelongue, Paris, France
- Germany (2):
  - University Hospital Heidelberg, Heidelberg
  - St. Franziskus Hospital, Münster
- Italy (4):
  - Azienda Ospedaliera Policlinico Sant'Orsola Malpighi, Bologna
  - Fondazione Poliambulanza, Brescia
  - Azienda Ospedaliero-Universitaria di Padova, Padua
  - Ospedale di Circolo e Fondazione Macchi, Varese
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - Erasmus Medical Center, Rotterdam
- Spain (2):
  - Hospital Universitario Central de Asturias (HUCA), Oviedo
  - University Hospital of Santiago de Compostela, Santiago de Compostela

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Usai MV, Gargiulo M, Haulon S, Tielliu I, Boeckler D, Verhagen H, Fernandez AM, Austermann MJ. One-year results of a balloon expandable endoprosthesis as a bridging stent for branched endovascular aortic repair. J Vasc Surg. 2023 Dec;78(6):1376-1382.e2. doi: 10.1016/j.jvs.2023.07.061. Epub 2023 Aug 11. PMID 37572891

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GORE VIABAHN VBX Balloon Expandable Endoprosthesis
Started | 280
Completed | 210
Not Completed | 70

BASELINE CHARACTERISTICS:
Arm/Group | GORE VIABAHN VBX Balloon Expandable Endoprosthesis
Number analyzed (Participants) | 280
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 68
  >=65 years | 212
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.7 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75
  Male | 205
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 60
  Italy | 77
  France | 8
  Germany | 92
  Spain | 43

OUTCOME MEASURES:

1. Primary Outcome: Composite of Procedural Success and Freedom From VBX Stent Graft-related Serious Adverse Events
Description: Number of study subjects experiencing Procedural Success and free from VBX Stent Graft-related Serious Adverse Events within 30 days of index procedure.
  Procedural Success is defined as: successful access, delivery, accurate deployment, and withdrawal of catheters with patent VBX Stent Graft at end of procedure.
Time Frame: 30 days post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | GORE VIABAHN VBX Balloon Expandable Endoprosthesis
Number analyzed (Participants) | 280
Participants | 274

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | GORE VIABAHN VBX Balloon Expandable Endoprosthesis
All-Cause Mortality (participants affected / at risk) | 49/280
Serious Adverse Events (participants affected / at risk) | 153/280
Other Adverse Events (participants affected / at risk) | 15/280
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GORE VIABAHN VBX Balloon Expandable Endoprosthesis (N=280)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Blood loss anemia (Blood and lymphatic system disorders) | 1 (1)
Macrocytic anemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Acute heart failure (Cardiac disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Acute myocardial infarction type 2 (Cardiac disorders) | 1 (1)
Aortic valve insufficiency (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Atrioventricular block (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2)
Cardiac asthma (Cardiac disorders) | 1 (1)
Cardiac ischaemia (Cardiac disorders) | 1 (1)
Cardiac ischemia (Cardiac disorders) | 1 (1)
Cardiac rupture (Cardiac disorders) | 1 (1)
Congestive heart failure (Cardiac disorders) | 3 (3)
Coronary heart disease (Cardiac disorders) | 1 (1)
Decompensation cardiac (Cardiac disorders) | 5 (5)
Heart failure (Cardiac disorders) | 3 (3)
Mitral valve insufficiency (Cardiac disorders) | 2 (2)
Myocardial infarction (Cardiac disorders) | 2 (3)
Non STEMI (Cardiac disorders) | 1 (1)
Right heart failure (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Abdominal wall hematoma (Gastrointestinal disorders) | 1 (1)
Bowel ischemia (Gastrointestinal disorders) | 1 (1)
Bowel obstruction (Gastrointestinal disorders) | 1 (1)
Celiac artery stenosis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Femoral hernia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1)
Hematochezia (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Intestinal polyp bleeding (Gastrointestinal disorders) | 1 (1)
Ischemic colitis (Gastrointestinal disorders) | 2 (2)
Mesenteric artery embolism (Gastrointestinal disorders) | 1 (1)
Mesenteric ischemia (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Proctorrhagia (Gastrointestinal disorders) | 1 (1)
Retroperitoneal hematoma (Gastrointestinal disorders) | 2 (2)
Splenic artery aneurysm (Gastrointestinal disorders) | 1 (1)
Arterial stent occlusion (General disorders) | 1 (1)
Death from natural causes (General disorders) | 1 (1)
Distal stent-induced new entry (General disorders) | 1 (1)
Extravasation of drug (General disorders) | 1 (1)
In-stent arterial restenosis (General disorders) | 4 (5)
In-stent arterial stenosis (General disorders) | 1 (1)
In-stent venous restenosis (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Multi organ failure (General disorders) | 1 (1)
Multiorgan failure (General disorders) | 1 (1)
Reduced general condition (General disorders) | 1 (1)
Renal stent-graft thrombosis (General disorders) | 1 (1)
Stent thrombosis (General disorders) | 2 (2)
Stent-graft endoleak type IA (General disorders) | 4 (4)
Stent-graft endoleak type IB (General disorders) | 4 (4)
Stent-graft endoleak type IC (General disorders) | 5 (5)
Stent-graft endoleak type II (General disorders) | 10 (12)
Stent-graft endoleak type III (General disorders) | 4 (5)
Stent-graft endoleak type IIIA (General disorders) | 1 (1)
Stent-graft stenosis (General disorders) | 2 (3)
Stent-graft thrombosis (General disorders) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 2 (2)
Unknown cause of death (General disorders) | 4 (4)
Wound healing disturbance of (General disorders) | 2 (3)
Acute cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Hepatic artery stenosis (Hepatobiliary disorders) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1)
Bacterial endocarditis (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3)
COVID-19 pneumonia (Infections and infestations) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Graft infection (Infections and infestations) | 1 (1)
Infected seroma (Infections and infestations) | 1 (1)
Infected toe (Infections and infestations) | 1 (1)
Meningitis (Infections and infestations) | 1 (1)
Necrotizing fasciitis (Infections and infestations) | 1 (1)
Pneumococcal sepsis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 8 (8)
Postoperative wound infection (Infections and infestations) | 1 (1)
Prosthesis related infection (Infections and infestations) | 1 (1)
Puncture site infection (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
SARS-CoV-2 infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 7 (7)
Septic shock (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3)
Urosepsis (Infections and infestations) | 2 (2)
Vascular stent infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 2 (2)
Arteriovenous fistula site stenosis (Injury, poisoning and procedural complications) | 1 (1)
Arteriovenous graft site stenosis (Injury, poisoning and procedural complications) | 2 (2)
False aneurysm (Injury, poisoning and procedural complications) | 2 (2)
Femoral artery pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture subtrochanteric (Injury, poisoning and procedural complications) | 1 (1)
Fractured ribs (Injury, poisoning and procedural complications) | 1 (1)
Postimplantation syndrome (Injury, poisoning and procedural complications) | 3 (3)
Postoperative hematoma (Injury, poisoning and procedural complications) | 2 (2)
Vascular access site occlusion (Injury, poisoning and procedural complications) | 2 (2)
Vascular access site thrombosis (Injury, poisoning and procedural complications) | 3 (9)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 4 (5)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 (1)
Wound bleeding (Injury, poisoning and procedural complications) | 2 (2)
Aspiration bronchial (Investigations) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Coxarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Gonarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Low back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Ameloblastic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cholangiocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gallbladder tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Kidney cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Metastatic breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anterior spinal artery syndrome (Nervous system disorders) | 3 (3)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Dural arteriovenous fistula (Nervous system disorders) | 1 (1)
Hemorrhagic stroke (Nervous system disorders) | 1 (1)
Ischemic stroke (Nervous system disorders) | 2 (3)
Middle cerebral artery stroke (Nervous system disorders) | 1 (1)
Spinal cord ischemia (Nervous system disorders) | 3 (3)
Stroke (Nervous system disorders) | 2 (2)
Transient ischemic attack (Nervous system disorders) | 1 (1)
Device dislocation (Product Issues) | 1 (1)
Device migration (Product Issues) | 1 (1)
Stent migration (Product Issues) | 1 (1)
Stent occlusion (Product Issues) | 8 (9)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Acute on chronic renal failure (Renal and urinary disorders) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 3 (3)
Acute renal insufficiency (Renal and urinary disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Renal artery dissection (Renal and urinary disorders) | 3 (3)
Renal artery occlusion (Renal and urinary disorders) | 4 (5)
Renal failure (Renal and urinary disorders) | 4 (4)
Renal function aggravated (Renal and urinary disorders) | 1 (1)
Renal insufficiency (Renal and urinary disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1)
Vaginal prolapse (Reproductive system and breast disorders) | 1 (1)
Acute pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Heel ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Hepatectomy (Surgical and medical procedures) | 1 (1)
Radical nephrectomy (Surgical and medical procedures) | 1 (1)
Aneurysm enlargement (Vascular disorders) | 1 (1)
Aneurysm of aortic arch (Vascular disorders) | 1 (1)
Aortic thrombosis (Vascular disorders) | 1 (1)
Arterial stenosis (Vascular disorders) | 1 (1)
Brachiocephalic vein stenosis (Vascular disorders) | 1 (2)
Femoral artery thrombosis (Vascular disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hypovolemic shock (Vascular disorders) | 1 (1)
Iliac artery aneurysm (Vascular disorders) | 1 (1)
Iliac artery occlusion (Vascular disorders) | 1 (1)
Iliac artery restenosis (Vascular disorders) | 1 (1)
Iliac artery stenosis (Vascular disorders) | 3 (3)
Iliac artery thrombosis (Vascular disorders) | 3 (4)
Limb ischemia (Vascular disorders) | 1 (1)
Lower limb ischemia (Vascular disorders) | 1 (1)
Lymphatic fistula (Vascular disorders) | 1 (1)
Peripheral arterial disease (Vascular disorders) | 1 (2)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease Fontaine stage III (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease Fontaine stage IIb (Vascular disorders) | 1 (1)
Phlebitis arm (Vascular disorders) | 1 (1)
Popliteal artery aneurysm (Vascular disorders) | 2 (3)
Subclavian artery thrombosis (Vascular disorders) | 1 (1)
Superficial femoral arterial stenosis (Vascular disorders) | 1 (2)
Superficial femoral artery occlusion (Vascular disorders) | 1 (1)
Thoracic aortic aneurysm (Vascular disorders) | 1 (1)
Thoracic aortic aneurysm enlargement (Vascular disorders) | 1 (1)
Type A aortic dissection (Vascular disorders) | 1 (1)
Type B aortic dissection (Vascular disorders) | 1 (1)
Vascular stenosis (Vascular disorders) | 1 (1)
Venous stenosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GORE VIABAHN VBX Balloon Expandable Endoprosthesis (N=280)
Stent-graft endoleak type II (General disorders) | 15 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-08): https://cdn.clinicaltrials.gov/large-docs/04/NCT03720704/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/04/NCT03720704/SAP_001.pdf